CLINICAL TRIAL: NCT05143216
Title: High Concentration Oxygen Therapy for Pneumocephalus After Evacuation of Chronic Subdural Haematoma: A Prospective Observational Study
Brief Title: High Concentration Oxygen Therapy for Pneumocephalus in Chronic Subdural Haematoma: A Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. David Yuen Chung CHAN (Other)
Responsible Party: Sponsor-Investigator, Dr. David Yuen Chung CHAN, Assistant Professor (Neurosurgery), Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: WON-20210111-18486
Record Dates: First submitted 2021-12-02; First posted 2021-12-03 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic subdural hematoma; Oxygen therapy
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic subdural haematoma post burr-hole drainage: Chronic subdural haematoma post burr-hole drainage
  Interventions: Other: Low concentration oxygen group: Room air (0-2Litre Oxygen via Nasal Canula); Other: High concentration oxygen group: Room air (12-15Litre Oxygen via Non-rebreather Mask)

INTERVENTIONS:
Other: Low concentration oxygen group: Room air (0-2Litre Oxygen via Nasal Canula) — Low concentration oxygen group: Room air (0-2Litre Oxygen via Nasal Cannula)
Other: High concentration oxygen group: Room air (12-15Litre Oxygen via Non-rebreather Mask) — High concentration oxygen group: Room air (12-15Litre Oxygen via Non-rebreather Mask)

SUMMARY:
Normobaric oxygen therapy was shown to be effective in reducing post craniotomy pneumocephalus. Theoretical assessment of normobaric oxygen therapy in treating pneumocephalus has shown that a higher level of oxygen concentration will significantly decrease the time for absorption of pneumocephalus. The therapeutic efficacy is not fully established in patients with chronic subdural hematoma after burr hole drainage. Both radiological outcomes and clinical outcomes would be evaluated.

DETAILED DESCRIPTION:
Chronic subdural hematoma (CSDH) is not a benign disease. Morbidity and mortalities were high especially in those with recurrence requiring reoperations. The use of subdural drain after burr hole drainage is an excellent example demonstrating that by reducing CSDH recurrence, a significant improvement in functional outcomes can be observed.

Pneumocephalus is very common after burr hole drainage for CSDH. The use of high-flow oxygen had been reported to be effective in small case series, showing effectiveness in clinical and radiological outcomes. However, no large, prospective, controlled trial has been conducted to establish the efficacy of oxygen therapy on functional outcomes for patients with pneumocephalus after burr hole drainage in CSDH.

Bilateral CSDH has a different prognosis and is associated with a poorer outcome.

In addition to treating pneumocephalus, the use of perioperative oxygen has been suggested to minimize tissue hypoxemia and infection. In a study published in the New England Journal of Medicine, the use of perioperative supplementary oxygen was shown to reduce surgical site infection.

Hyperoxia with oxygen therapy has shown to be safe with minimal changes to the cerebral blood flow (CBF) from functional magnetic resonance imaging (fMRI).

Research Questions

1. Does post-operative high-flow oxygen improve pneumocephalus in terms of volume reduction in CSDH patients after burr-hole drainage?
2. Does post-operative high-flow oxygen reduce the recurrence rate of CSDH (radiologically) if pneumocephalus volume is reduced after oxygen therapy?
3. Does post-operative high-flow oxygen reduce the recurrence rate of CSDH (clinically), as defined by symptomatic recurrence requiring reoperation, if pneumocephalus volume is reduced after oxygen therapy?
4. Does post-operative high-flow oxygen improve CSDH patients' functional outcome in terms of modified Rankin Scale (mRS) at 3 months and 6 months? Hypothesis Oxygen therapy for CSDH patients with post-operative pneumocephalus will experience significant resorption of intracranial air within 24 hours. There is a reduction in recurrence rate in terms of the re-operation rates. There is an improvement in functional outcome in terms of mRS.

Aim of the Study To evaluate changes in pneumocephalus volume and functional outcome after oxygen therapy in post-operative CSDH patients treated by burr hole drainage, as compared to the standard care by breathing in room air or low concentration oxygen during the post-operative period.

Study Design Prospective randomized 1:1 parallel-arm study Methods and Randomization Patients will be recruited when they are considered fit for oxygen therapy as determined by the treating clinician. The timing of burr hole evacuation may vary according to the availability of the emergency operative time slot. The index intervention is postoperative oxygen therapy: 100% normobaric oxygen through a nonrebreather mask (NRM) at 12-15 Litre/minute consecutively for 24 hours. Removal of the nonrebreather mask is allowed during meals or other activities such as physiotherapy. The duration of mask removal would be documented. Compliance with NRM is considered to be good if the mask is kept > 90% of the time during the 24 hours treatment period. The reference intervention is standard post-operative care: the patient would be breathing in normobaric room air. For the reference arm, if the patient has desaturation (i.e. SaO2 < 93%), supplemental O2 therapy can be given to keep SaO2 > 93%. Arterial blood gas would be obtained by the clinicians when deemed necessary. If there is a significant deviation from the study protocol occurs, the patients will be analyzed according to their originally assigned groups (intention-to-treat principle).

Non-rebreather masks, when they are tightly applied, are associated with a lower aerosol dispersion distance (as compared to non-invasive positive pressure ventilation or venturi masks).

Interim data analysis would be performed and the study would be terminated if a significant difference in the primary outcome is observed.

ELIGIBILITY:
Inclusion Criteria:

Age greater than or equal to 18 years-old. Presence of chronic subdural haematoma (CSDH) as diagnosed radiologically either by computed tomography (CT) brain scan or magnetic resonance imaging (MRI).

Treatment of CSDH by burr-hole evacuation. Post operative pneumocephalus, as evidenced from post-operative CT Brain or MRI brain.

Negative test to SARS-nCoV-2, as evidenced by either deep throat saliva rapid test, deep throat saliva PCR test, nasopharyngeal swab real-time PCR test, or nasopharyngeal swab rapid test within seven days.

Exclusion Criteria:

Presence of pre-existing respiratory conditions such as chronic obstructive pulmonary disease (COPD) and hence not suitable for oxygen therapy.

Any pre-existing illness that renders the patient moderately or severely disabled before diagnosis with CSDH, such as a history of central nervous system infection.

CSDH arising from secondary causes, such as intracranial hypotension, thrombocytopenia, etc.

Any evidence or suspicion that there is communication between the pneumocephalus with the air cells (e.g. such as mastoid air cells) or air sinuses (e.g. frontal sinus).

Patients that need an additional procedure e.g. epidural blood patch, etc. Complications arising from the burr-hole operation or subdural drain insertion such as hemorrhage or surgical site infection requiring surgical intervention or deemed to affect the patient's long-term functional outcome.

Patients already on long-term steroid for pre-existing medical conditions. Patients who received instillation of subdural urokinase or tissue plasminogen activator via the subdural catheter(s).

Participation in other clinical trials within four weeks upon recruitment. Pregnancy or on breastfeeding. Any other reasons that the researchers consider the patients to be unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic subdural haematoma
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in pneumocephalus volume | 24 hours
  Changes in pneumocephalus volume
Changes in pneumocephalus volume | 48-72h hours
  Changes in pneumocephalus volume
Recurrence | 6 month

SECONDARY OUTCOMES:
Modified Rankins Scale | 3 month, 6 month

CONTACTS AND LOCATIONS:
Overall Officials: David YC CHAN, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Division of Neurosurgery, Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided